CLINICAL TRIAL: NCT06621030
Title: Evaluation of Correlations Between Volatile Organic Compounds (VOCs) Spectra Measured With GC-IMS and MOx-sensors and Venous Blood Glucose in Subjects With Type 2 Diabetes
Brief Title: Evaluation of Correlations Between Volatile Organic Compounds and Venous Blood Glucose in Subjects With Type 2 Diabetes
Acronym: Evo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BOYDSENSE (Industry)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); DCB Research AG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Evo Study
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
Keywords: Volatile Organic Compounds; Gas Chromatography - Ion Mobility Spectrometry; Rates of change of glucose values; Breath-analysis; Hyperglycaemia; Hypoglycaemia; Glucose excursions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: The intervention consists of inducing different glycaemic states in people with diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Exposure to various glycaemic states at different rates of change by administering glucose solution, insulin, or a standardized meal.
  Interventions: Device: MIB Breath Analyzer

INTERVENTIONS:
Device: MIB Breath Analyzer — Going through visit-specific blood glucose excursions by the administration of glucose and insulin (clamp), monitoring physiological processes, and measuring reference blood glucose values and VOC measurements in the breath using a GC IMS and the MIBs (investigational devices). Going through visit-specific blood glucose excursions by consuming a standardized meal, monitoring physiological processes, and measuring reference blood glucose values and VOC measurements in the breath using a GC-IMS and the MIBs (investigational devices) Imitating the glucose excursion from the meal excursion by infusing glucose and insulin (clamp), monitoring physiological processes, and measuring reference blood glucose values and VOC measurements in the breath using a GC-IMS and the MIBs (investigational devices).

SUMMARY:
The goal of this study is to evaluate correlations between VOCs in the breath and venous blood glucose values in various glycaemic states in people living with Type 2 Diabetes. VOCs are measured with a gold-standard GC-IMS device and a prototype of a novel breath analyzer. Participants will be exposed to different blood glucose levels at different rates of change by administering glucose solution and insulin and by a meal challenge.

DETAILED DESCRIPTION:
The research project aims to expand the understanding of correlations between VOCs in the breath and venous blood glucose levels in non-insulin-dependent people with Type 2 Diabetes. To better understand correlations, the subjects are exposed to hyperglycaemic, euglycaemic and hyposglcycaemic states at different rates of change by applying a hand clamp procedure, and the VOCs are compared after a standardized meal and the same excursion by applying a hand clamp procedure. Inter- and intraparticipant variability as well as the timing of changes in the VOC spectra compared to changes in the glucose values are of interest. Secondarily, the feasibility of estimating glycaemic states with a prototype of a novel breath analyzer is being investigated.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* T2D treated with one or more oral anti-diabetic drugs (incl GLP-1 and/or GIP)
* 10 years since T2D diagnosis
* HbA1c ≤8% (HbA1c based on last measurement by treating physician but not older than 120 days)
* Willingness to undergo study procedures
* Age 45 -70 years (inclusive)

Exclusion Criteria:

* Pregnancy and/or lactation period
* Currently on chronic or occasional treatment with pulmonary drugs
* Insulin dependency
* Smoking (last cigarette within the last six months)
* BMI above 30 kg/m²
* Lp(a) above 125 nmol/l
* LDL not in the individual target range of an earlier cholesterol goal according ESC guideline 2021 (LDL based on last measurement by treating physician but not older than 30 days)
* Irregular 12-lead ECG or increased carotid plaque burden based on a three-point sonography. Both examinations are performed and evaluated according to the investigator's judgment.
* History of, or manifested, cardiovascular diseases
* Medical history of epilepsy or other neurological disease associated with seizure events
* Known sensitivity to medical grade adhesives
* Comorbidities that are suspected to alter the VOC spectra
* Participation in another investigation with an investigational drug within the 30 days preceding and during the present investigation
* Not able to understand, write or read German

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
VOC spectra | 6-8 hour study visit
  Primary outcome focuses on VOC spectra (measured with the GC-IMS) across varying intravenous blood glucose levels

SECONDARY OUTCOMES:
Inter-Participant VOC Variability | 6-8 hour study visit
  Evaluation of VOC spectral differences measured with the GC-IMS among participants under identical glycemic states.
Intra-Participant VOC Variability | 6-8 hour study visit
  Comparison of VOC spectral differences measured with the GC-IMS within the same participant across different glycemic states.
MIB VOC Spectra Analysis | 6-8 hour study visit
  Investigation of VOC spectra (measured with the MIB) in diverse intravenously measured glycemic states.
VOC Spectra Response Time | 6-8 hour study visit
  Assessment of the delay in VOC spectral shifts relative to changes in venous glucose from fluctuating to stable states at different change rates.
Comparison of meal vs clamp induced VOC changes | 6-8 hour study visit
  Analysis of VOC spectral differences between natural post-meal glucose increases and clamp-induced glucose elevations measured with the GC-IMS.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Flacke, Dr, Study Chair — BOYDSense SAS; Markus Laimer, Prof, Principal Investigator — Universitätsklinik für Diabetologie, Endokrinologie, Ernährungsmedizin & Metabolismus (UDEM)

IPD SHARING:
Plan to Share IPD: No